CLINICAL TRIAL: NCT05373836
Title: Relationship of PNI and Clinical Outcome in Patients Undergoing Brain Tumor Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, PhD, Clinical Associate Professor, Seoul National University Hospital
Other Study IDs: PNI_Brain tumor
Record Dates: First submitted 2022-04-24; First posted 2022-05-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Clinical Outcome
Keywords: nutritional index; brain tumor surgery; mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- brain tumor surgery: adult patients undergoing brain tumor surgery
  Interventions: Diagnostic Test: prognostic nutritional index calculated from laboratory parameters

INTERVENTIONS:
Diagnostic Test: prognostic nutritional index calculated from laboratory parameters — Calculated nutritional index using laboratory results of serum albumin, lymphocyte count, and cholesterol

SUMMARY:
There are several predictors of clinical outcome in patients undergoing brain tumor surgery. Among those, nutritional parameters and calculated nutritional index are known to have ability to predict mortality and clinical outcomes in some patients with brain tumor. However, there are lack of consistent results on predictability of nutritional index and clinical outcome in patients undergoing brain tumor surgery.

DETAILED DESCRIPTION:
In this retrospective study, we evaluated the relationship between prognostic nutritional index, which was calculated from laboratory parameters, and clinical outcome including mortality in patients undergoing brain tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing brain tumor surgery at Seoul National University Hospital, South Korea

Exclusion Criteria:

* Lack of results of laboratory parameters, such as serum albumin, lymphocyte count, cholesterol
* Lack of data on clinical outcome, including mortality, acute kidney injury, renal replacement therapy, length of hospital stay, and other major adverse outcome

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing brain tumor surgery at Seoul National University Hospital, South Korea
Sampling Method: Non-Probability Sample
Enrollment: 3263 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
predictability of prognostic nutritional index for mortality after brain tumor surgery | From date of surgery until the date of death from any cause, whichever came first, assessed up to 50 years
  Odds ratio of prognostic nutritional index for postoperative mortality

SECONDARY OUTCOMES:
predictability of prognostic nutritional index for acute kidney injury after brain tumor surgery | From date of surgery until the date of acute kidney injury from any cause, whichever came first, assessed up to 50 years
  Odds ratio of prognostic nutritional index for postoperative acute kidney injury
predictability of prognostic nutritional index for renal replacement therapy after brain tumor surgery | From date of surgery until the date of renal replacement therapy from any cause, whichever came first, assessed up to 50 years
  Odds ratio of prognostic nutritional index for postoperative renal replacement therapy
relationship of prognostic nutritional index for length of hospital stay after brain tumor surgery | From date of surgery until the date of hospital discharge
  Odds ratio of prognostic nutritional index for length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided